CLINICAL TRIAL: NCT01774136
Title: The Effectiveness of an HIV-adapted IMCI Training and Supervision Programme of Community Caregivers to Support Interventions That Will Reduce MTCT and Improve Delivery of Other Essential Newborn and Child Survival Interventions
Brief Title: Effectiveness of an HIV-adapted IMCI Training and Supervision Programme for Community Health Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); World Health Organization (Other); Institute for Healthcare Improvement (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Dr. Jennifer Reddy, Director, University of KwaZulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nompilo
Record Dates: First submitted 2013-01-20; First posted 2013-01-23 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Prevention of Mother-to-child Transmission of HIV; Antenatal Health Care Utilization; Postnatal Health Care Utilization; Infant Feeding Practices
Keywords: community health workers; HIV; PMTCT; antenatal; postnatal; breastfeeding; South Africa
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced HIV and MCH training for CHW (Experimental): The intervention includes two components: (1) a 2-week HIV/C-IMCI training for CCGs and their associated facilitators and supervisors, and (2) continuous support and supervision following the continuous quality improvement (CQI) framework, a low-technology approach to management and supervision of health programs.
  Interventions: Behavioral: Enhanced HIV and MCH training for CHW
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Enhanced HIV and MCH training for CHW
  Arms: Enhanced HIV and MCH training for CHW

SUMMARY:
This is a cluster randomized controlled trial (C-RCT) to evaluate the effectiveness of a Community-Integrated Management of Childhood Illness (C-IMCI) training for community caregivers (CCGs), adapted to include HIV-related interventions, on the delivery of maternal, newborn and child health interventions within households in rural communities in Ugu District, KwaZulu-Natal (KZN) Province, South Africa. The intervention includes two components: (1) a 2-week HIV/C-IMCI training for CCGs and their associated facilitators and supervisors, and (2) continuous support and supervision following the continuous quality improvement (CQI) framework, a low-technology approach to management and supervision of health programs. The primary objectives of the proposed evaluation are to measure the effect of the intervention on key outcomes, including early uptake of antenatal care, facility based delivery, postnatal visits, coverage of exclusive breastfeeding, and uptake of HIV PCR testing in infants at 6 weeks. We will also examine the effects of the intervention on immunization uptake up to 12 months and knowledge and practices of CCGs and mothers pertaining to maternal, newborn and child health.

ELIGIBILITY:
Inclusion Criteria:

Community caregivers

* CCGs who work in Ugu District
* age 18 years or older
* with grade 9 education or greater

Mothers

* Mothers age 18 years and older who delivered a live-born infant within the prior 12 months
* Reside in households served by participating CCGs.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1342 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of antenatal booking before 20 weeks gestation | 1 year
Prevalence of presentation for post-natal care within 7 days of delivery | 1 year
Prevalence of exclusive breast-feeding practice at 14 weeks | 1 year
Coverage of HIV PCR testing at 6 weeks | 1 year

SECONDARY OUTCOMES:
Proportion of women who attended for antenatal care at least 4 times in pregnancy | 1 year
Proportion of deliveries by skilled birth attendant at a health facility | 1 year
Proportion of age-eligible infants who received recommended immunizations at 6, 10, and 14 weeks and 9 and 12 months | 1 year
Proportion of children whose growth was monitored by CCG at home | 1 year
Prevalence of exclusive breast-feeding practice at 6 months | 1 year
Proportion of women without known HIV-positive status who received HIV test in pregnancy | 1 year
Proportion of women without known HIV-positive status who received HIV test result in pregnancy | 1 year
Proportion of HIV-positive women who received CD4 test results | 1 year
Proportion of HIV-positive women who received ARV prophylaxis in pregnancy and during delivery | 1 year
Proportion of infants born to HIV-positive mothers who received ARV prophylaxis following birth (including during breastfeeding where appropriate) | 1 year
Knowledge and practices of mothers in the community regarding: infant feeding, HIV, availability of interventions to reduce HIV transmission, newborn care practices and recognition of serious illness in children and management of childhood illnesses | 1 year
Knowledge and practices of CCGs with regards to: HIV-specific interventions to improve maternal health, reduce HIV transmission and improve child survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reddy, MBChB, Principal Investigator — 20,000+ Partnership, University of KwaZulu-Natal
Locations (1):
- 20000+ Partnership, UKZN, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Horwood C, Butler L, Barker P, Phakathi S, Haskins L, Grant M, Mntambo N, Rollins N. A continuous quality improvement intervention to improve the effectiveness of community health workers providing care to mothers and children: a cluster randomised controlled trial in South Africa. Hum Resour Health. 2017 Jun 13;15(1):39. doi: 10.1186/s12960-017-0210-7. PMID 28610590